CLINICAL TRIAL: NCT02667379
Title: Evaluation of Skin Prick Tests in Cat Allergic Patients With Cat Dander Samples Obtained Before and After Vaccinating the Cat
Brief Title: Skin Tests in Cat Allergic Patients With Cat Dander Samples Obtained Before and After Vaccinating the Cat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ZU-HypoCat-001
Record Dates: First submitted 2016-01-20; First posted 2016-01-28 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Hypersensitivity
Keywords: Cat; allergy; dander; Fel d 1; Felis domesticus
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic skin testing (Other): Diagnostic skin testing with cat dander samples on volar forearms.
  Interventions: Other: Diagnostic skin testing

INTERVENTIONS:
Other: Diagnostic skin testing — 14 Skin prick tests on each volar forearm with cat dander samples.

SUMMARY:
Determination of allergenicity of cat dander samples obtained before and after vaccinating the cat

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Male or female between 18 years to 65 years
* Confirmed cat allergy (positive skin prick test)

Exclusion Criteria:

* Diseases or medications, influencing the skin tests or impairing the correct conduct and evaluation of the study
* History of anaphylactic reaction
* Pregnancy
* Skin irritations in test area
* Participation in another clinical trial within the last 30 days and during the present study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Wheal size of allergic skin reaction in mm² measured 15 minutes after application of test substance | 15 minutes
  The primary variable will be the wheal size area of the immediate phase reaction in mm² measured after 15 minutes. Determination of the concentration threshold at which no more skin reactivity can be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kuendig, MD, Principal Investigator — University Hospital Zurich, Dept Dermatology
Locations (1):
- University Hospital Zurich, Dept of Dermatology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No